CLINICAL TRIAL: NCT04519814
Title: A Prospective, Multicenter Clinical Investigation to Evaluate Safety and Effectiveness of VISULAS Green Selective Laser Trabeculoplasty (SLT)
Brief Title: Safety and Effectiveness of VISULAS Green Selective Laser Trabeculoplasty (SLT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1703PM
Record Dates: First submitted 2020-07-22; First posted 2020-08-20 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Primary Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- all eligible patients (Experimental): A total of 40 eyes in 40 consecutive patients, 22 years of age or older, with primary open-angle glaucoma (HPG + NPG), who did not reach target pressure, agree to participate in the study, and will be able to complete clinical follow-up and evaluation.
  Interventions: Procedure: selective laser trabeculoplasty (SLT)

INTERVENTIONS:
Procedure: selective laser trabeculoplasty (SLT) — Treatment will be performed on Day 0 using the VISULAS green with Option CSLT for SLT treatment and a mirror goniolens to visualize the trabecular meshwork. The initial energy level is set according to the grade of angle pigmentation and bubble formation. Approximately one hundred non-overlapping lesions will be applied in a single session to 360° of the trabecular meshwork.

SUMMARY:
An interventional, open, prospective, multi-center pre-market clinical investigation according to §§20-23a Medizinproduktegesetz (MPG, medical devices act), in which a total of 40 eyes of 40 consecutive patients at up to five (5) clinical sites will be enrolled, treated with the VISULAS green with option CSLT, and followed for a three months period.

The primary objective of this clinical investigation is to evaluate safety and effectiveness of SLT with the VISULAS green laser with option CSLT.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 22 years of age or older, primary open-angle glaucoma (HPG + NPG), who did not reach target pressure .
* IOP with or without medications ≥17 mmHg in the study eye
* Chamber angle Shaffer 3 and 4
* Patients must be legally competent and able to give consent and must have read, understood and signed patient information leaflet and consent to undergo SLT in one eye
* Patients are willing and able to return for follow-up examinations
* In the opinion of the investigator, the patient will be compliant and have a high probability of completing the clinical investigation and all required procedures

Exclusion Criteria:

* Corneal disease or pathology in a way that distortion of laser light in the study eye can be expected or that precludes stabilization of the cornea by the contact glass, visibility of the trabecular meshwork or transmission of laser wavelength
* Strong clouding of the anterior ocular media (e.g. the lens due to dense cataract) and the vitreous body (e.g. due to strong vitreous hemorrhage) in either eye
* Deep orbits and/or narrow palpebral fissures
* Corneal or conjunctival abnormality precluding contact lens adaptation in either eye
* History of Amblyopia in either eye
* Any contraindications to SLT in study eye.
* Any kind of planned ocular surgeries during the next 3 months (for example, cataract surgery) in either eye
* Previous intraocular or corneal surgery of any kind (except cataract surgery longer than three months prior to the clinical investigation), including surgical glaucoma intervention in study eye before the clinical investigation.
* Signs of Fuchs' Dystrophy (e.g. corneal endothelial guttata) in either eye
* Active or history of Uveitis in either eye
* Congenital glaucoma in either eye
* Diabetic retinopathy or branch retinal vein occlusion with the risk to develop neovascularizations in either eye
* Heavily pigmented trabecular meshwork due to pseudoexfoliation syndrome or pigment dispersion glaucoma in either eye
* Degenerative disorders of the central nervous system if it prevents proper compliance or the ability to undergo the tests in the clinical investigation (e.g. Parkinson Disease, Alzheimer Disease, or other forms of dementia)
* History of or has a current, clinically significant major psychiatric disorder (e.g., major depressive disorder, psychosis, schizophrenia)
* Patients who are pregnant, lactating, or of child-bearing potential and not practicing a medically approved method of birth control.
* Enrollment in another drug or device study within the prior 3 months

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
mean absolute change in intraocular pressure (IOP) compared to baseline at month 1 | one (1) month
  The endpoint is the mean change in IOP (Absolute value, mmHg) of the study cohort compared to baseline at month 1

SECONDARY OUTCOMES:
mean relative change in intraocular pressure (IOP) compared to baseline at month 1 | one (1) month
  The endpoint is the mean change in IOP (relative value, %) of the study cohort compared to baseline at month 1
mean absolute change in intraocular pressure (IOP) compared to baseline at month 3 | three (3) months
  The endpoint is the mean change in IOP (Absolute value, mmHg) of the study cohort compared to baseline at month 3
mean relative change in intraocular pressure (IOP) compared to baseline at month 3 | three (3) months
  The endpoint is the mean change in IOP (relative value, %) of the study cohort compared to baseline at month 3

OTHER OUTCOMES:
rate of patients achieving >0 to <10% IOP reduction from baseline | three (3) month
  The following exploratory endpoint will be determined additionally:
  - rate of patients achieving >0 to <10% IOP reduction from baseline at 1 and 3 months
rate of patients achieving 10% to <20% IOP reduction from baseline | three (3) month
  The following exploratory endpoint will be determined additionally:
  - rate of patients achieving 10% to <20% IOP reduction from baseline at 1 and 3 months
rate of patients achieving ≥20% IOP reduction from baseline | three (3) month
  The following exploratory endpoints will be determined additionally:
  - rate of patients achieving ≥20% IOP reduction from baseline at 1 and 3 months.
Post-operative intraocular pressure (IOP) in mmHg | one (1) day
  Outcome Parameters Safety: Post-operative intraocular pressure (IOP) in mmHg: 1h, 1d
Rate of intraoperative Adverse Device Effects | one (1) day
  Outcome Parameters Safety: Rate of intraoperative Adverse Device Effects
Rate of Adverse Device Effects and Device Deficiencies | three (3) month
  Outcome Parameters Safety: Rate of Adverse Device Effects and Device Deficiencies over the entire course of the investigation
Rate of Adverse Events and Severe Adverse Events | three (3) month
  Outcome Parameters Safety: Rate of Adverse Events and Severe Adverse Events over the entire course of the clinical investigation

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Klinik und Poliklinik für Augenheilkunde, TU Dresden, Dresden
  - Internationale Innovative Ophthalmochirurgie GbR, Düsseldorf
  - Augenarztpraxis am Dreiecksplatz, Kiel, Kiel
  - Klinik für Augenheilkunde, UK Schleswig Holstein, Kiel
  - Augentagesklinik Rheine, Rheine

REFERENCES:
- [Background] Pillunat KR, Kretz FTA, Koinzer S, Ehlken C, Pillunat LE, Klabe K. Effectiveness and safety of VISULAS(R) green selective laser trabeculoplasty: a prospective, interventional multicenter clinical investigation. Int Ophthalmol. 2023 Jul;43(7):2215-2224. doi: 10.1007/s10792-022-02617-7. Epub 2022 Dec 26. PMID 36572747